CLINICAL TRIAL: NCT00860613
Title: Medical Nutrition Therapy Program for Pregnant Women With Diabetes: Evaluation of Two Different Dietary Strategies on Metabolic Control, Maternal and Fetal Nutritional Status and Cost Effectiveness.
Brief Title: Medical Nutrition Therapy Program for Pregnant Women With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Perinatologia Isidro Espinosa de los Reyes (Other Government)
Responsible Party: Otilia Perichart Perera, Instituto Nacional de Perinatologia Isidro Espinosa de los Reyes
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 212250-02091
Record Dates: First submitted 2009-03-11; First posted 2009-03-12 (Estimated); Last update posted 2009-03-12 (Estimated); Status verified 2009-03

CONDITIONS: Gestational Diabetes; Type 2 Diabetes
Keywords: gestational diabetes; medical nutrition therapy program; glucose monitoring; metabolic control; nutritional status; cost effectiveness
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): women in this group received usual medical treatment and counseling from a nutritionist and diabetes educator. They received a specific diet using carbohydrate counting (40-45% of carbohydrates)and a moderate energy restriction. Weight gain, adequacy of diet, results of the self glucose monitoring, and ketonuria were evaluated every two weeks. They also received education on diabetes, diet and glucose monitoring.
  Interventions: Other: medical nutrition therapy program
- 2 (Experimental): Women in this group received usual medical treatment and counseling from a nutritionist and diabetes educator. The diet they received was based on carbohydrate counting (40-45% of carbohydrates), but recommended only low-moderate glycemic index foods. Weight gain, adequacy of diet, results of the self glucose monitoring, and ketonuria were evaluated every two weeks. They also received education on diabetes, diet and glucose monitoring.
  Interventions: Other: medical nutrition therapy program
- 3 (No Intervention): women in this group received the current hospital treatment. They did not receive any intervention except for the self glucose monitoring that they did every two weeks. Weight gain and the results of the self glucose monitoring, were evaluated every two weeks.

INTERVENTIONS:
Other: medical nutrition therapy program — the dietary guidelines were based on the Nutrition Practice guidelines for gestational diabetes developed by the American Dietetic Association. Dietary strategies were based on carbohydrate counting and/or restriction of high glycemic index foods. Even carbohydrate distribution throughout the day was emphasized.
  Arms: 1; 2

SUMMARY:
No dietary strategies have been designed and proved for Mexican pregnant women with diabetes. This is a randomized clinical trial of pregnant women with pregestational type 2 diabetes and gestational diabetes that were followed every two weeks until labor to assess the impact of the MNT program on metabolic control, maternal and fetal nutritional status and cost effectiveness. Participants were randomly assigned to one of three medical nutrition therapy (MNT) groups: the MNT 1 group (n=38) received usual medical treatment, counseling from a nutritionist and diabetes educator, using carbohydrate counting (40-45% of carbohydrates)with an intensive educational component; MNT2 group (n=50) had the same treatment, but included only low-moderate glycemic index foods; and NO-MNT group (n=45) received the current hospital treatment. All women will receive a glucose meter so they do self glucose monitoring (pre and postprandial) 2 times a weeks 6 times a day. Weight gain, dietary consumption and glucose concentrations will be evaluated every two weeks. Fetal outcomes (weight, length and presence of complications)will be measured at labor.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with gestational diabetes (Freinkle´s classification: type A2 and B1) or pregestational type 2 diabetes.
* less than 30 weeks of gestation
* women who plan to attend their pregnancy at the institution (INPerIER)

Exclusion Criteria:

* women with type 1 pregestational diabetes or gestational diabetes type A1.
* women with multiple pregnancies
* women with renal or hepatic disease
* women who could not follow the dietary recommendations within the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 162 (Actual)
Dates: Start 2004-02; Primary Completion 2007-06 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
metabolic control | every two weeks

SECONDARY OUTCOMES:
maternal nutritional status | every two weeks
fetal nutritional status | at labor
cost effectiveness | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Vadillo-Ortega, M.D, PhD, Study Chair — Instituto Nacional de Perinatología Isidro Espionosa de los Reyes; Otilia Perichart-Perera, M.S, RD, Principal Investigator — Instituto Nacional de Perinatología Isidro Espionosa de los Reyes; Margie Balas-Nakash, B.S, Study Chair — Instituto Nacional de Perinatología Isidro Espionosa de los Reyes; Adalberto Parra-Covarrubias, M.D, Study Chair — Instituto Nacional de Perinatologia Isidro Espinosa de los Reyes; Ameyalli Rodriguez-Cano, B.S, Study Chair — Instituto Nacional de Perinatología Isidro Espinosa de los Reyes
Locations (1):
- Instituto Nacional de Perinatologia Isidro Espinosa de los Reyes, Mexico City, Mexico City, Mexico